CLINICAL TRIAL: NCT03198169
Title: 2-part, Randomized, Double Blind, Prospective, Single Center, Controlled Trial to Investigate an Antimicrobial Skin and Wound Cleanser and an Antimicrobial Barrier Film Dressing on the Rates of Healing for Chronic Wounds
Brief Title: A Study to Investigate Two Atteris Antimicrobial Products on Chronic Wound Healing.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inconsistent results in pilot phase
Sponsor: Atteris Healthcare, LLC (Industry)
Collaborators: Rochal Industries LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2017-07

CONDITIONS: Chronic Wounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active product containers and placebo product containers will have identical labels. Product numbers to differentiate active versus placebo will be assigned and known only by the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Active AWC + Active ABFD (Experimental): Active Antimicrobial Wound Cleanser + Active Antimicrobial Barrier Film Dressing + SOC
  Interventions: Device: Atteris Antimicrobial Skin and Wound Cleanser; Device: Atteris Antimicrobial Barrier Film Dressing
- Active AWC + Placebo ABFD (Experimental): Active Antimicrobial Wound Cleanser + Placebo Antimicrobial Barrier Film Dressing + SOC
  Interventions: Device: Atteris Antimicrobial Skin and Wound Cleanser; Device: Atteris Antimicrobial Barrier Film Dressing
- Placebo AWC + Active ABFD (Experimental): Placebo Antimicrobial Wound Cleanser + Active Antimicrobial Barrier Film Dressing + SOC
  Interventions: Device: Atteris Antimicrobial Skin and Wound Cleanser; Device: Atteris Antimicrobial Barrier Film Dressing
- Placebo AWC + Placebo ABFD (Experimental): Placebo Antimicrobial Wound Cleanser + Placebo Antimicrobial Barrier Film Dressing + SOC
  Interventions: Device: Atteris Antimicrobial Skin and Wound Cleanser; Device: Atteris Antimicrobial Barrier Film Dressing

INTERVENTIONS:
Device: Atteris Antimicrobial Skin and Wound Cleanser — Wounds will be cleansed with either the experimental wound cleanser or a placebo and will then be covered with standard of care wound dressings.
Device: Atteris Antimicrobial Barrier Film Dressing — Wounds will be covered with either the experimental barrier film dressing or a placebo and will then be covered with standard of care wound dressings.

SUMMARY:
This is a 2-part pilot study to determine the clinical effectiveness of two new antimicrobial products on the complete healing of chronic wounds.

DETAILED DESCRIPTION:
Part 1 of this study will involve 5 patients with qualified chronic wounds which will receive active treatment with both the Atteris Antimicrobial Skin and Wound Cleanser (AWC) and the Atteris Antimicrobial Barrier Film Dressing (ABFD) for a 6-week period with a 12 week follow-up in order to optimize the final study application protocols. Part 2 of this study is a randomized, double blind, 2 by 2 factorial, controlled study comparing the AWC and/or the ABFD with 100 research subjects and n=25 subjects per cell. Patients will be randomized to receive either active AWC and active ABFD, or active AWD and placebo ABFD, or placebo AWC and active ABFC, or AWC placebo and ABFD placebo in addition to standard of care (SOC). The active AWC active ABFD versus AWC placebo ABFD placebo statistical contrast will be of most importance and the clinical expectation is wounds treated with the active forms of these products will heal faster than wounds treated with double placebo and this will additionally provide data to power a future definitive study to compare the healing potential of the two therapeutic modalities (AWC, ABFD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 89
2. If IDDM or NIDDM, glycosylated hemoglobin, HgbA1c, ≤10%
3. Presence of chronic Wound of any etiology between 0.5 cm2 and 15 cm2, inclusive, post debridement
4. Wound has been present for at least 4 weeks, but not greater than 52 weeks at time of screening
5. Non-surgical wounds which meet the clinical definition of chronic between 0.5 cm2 and 15 cm2
6. Adequate arterial perfusion of the affected limb, defined as at least one of the following:

   1. Ankle-brachial index (ABI) ≥0.7 and ≤1.2
   2. Dorsum transcutaneous oxygen test ≥ 30 mm Hg
   3. Biphasic or triphasic Doppler waveforms at screening
7. Patient and/or caregiver have the ability and willingness to understand and comply with study procedures and give written, informed consent prior to enrollment in the study or initiation of study procedures.

Exclusion Criteria:

1. Suspected or confirmed signs/symptoms of active wound infection or gangrene
2. Hyperbaric Oxygen Therapy, any duration, within the past 12 months
3. Osteomyelitis
4. Use of oral or IV antibiotic/antimicrobial agents within 2 days (48 hours) of baseline
5. Subjects who have received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin,) within 28 days of screening
6. Subjects who have received dermal substitutes (e.g. Integra, collagen, micronized cadaver skin, bilayered cell therapy, dermal substitute, extracellular matrix etc.) within 28 days of screening.
7. Pyoderma gangrenosum, or Reynaud's disease
8. Wound with necrotic tissue covered with slough or eschar that cannot be debrided
9. Chronic wounds with exposed bone
10. Wounds with fistulas or deep sinus tracks of unknown depth
11. Active Charcot foot on the study limb
12. Receiving hemodialysis or peritoneal dialysis
13. History of malignancy excluding non-melanoma skin cancer
14. Treatment with radiation or chemotherapy within 3 months of screening
15. Known immunosuppression, excluding diabetes mellitus
16. Receiving (within 30 days of enrollment) or scheduled to receive a medication or treatment which is known to affect wound healing, such as systemic steroids (such as daily prednisone), immunosuppressive therapy, radiation or chemotherapy of any kind, autoimmune disease therapy or cytostatic therapy
17. Subjects with known alcohol or substance abuse within 6 months of screening
18. Subjects with known allergy to PHMB, acrylate polymer and silicone
19. Pregnancy or breastfeeding at time of screening
20. Participation in another investigational device, drug, or biological trial that may interfere with results within 6 months of screening

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Complete Closure | 6 weeks of active treatment
  Did the chronic wounds achieve complete closure as defined by 100% epithelialization requiring no additional treatment? (YES or NO)

SECONDARY OUTCOMES:
Infective episodes | 6 weeks
  The number of infective episodes for which oral or IV antibiotics are prescribed
Pain | 6 weeks
  Pain as reported using a Wong Baker Scale
Wound Dimension Decreases | 6 and 12 weeks
  The percentage change in wound size relative to the baseline measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Niezgoda, MD, FACHM, MAPWCA, CHWS, Principal Investigator — AZH Wound & Hyperbaric Center
Locations (1):
- AZH Wound & Hyperbaric Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] Gottrup F. A specialized wound-healing center concept: importance of a multidisciplinary department structure and surgical treatment facilities in the treatment of chronic wounds. Am J Surg. 2004 May;187(5A):38S-43S. doi: 10.1016/S0002-9610(03)00303-9. PMID 15147991
- [Background] Wicke C, Bachinger A, Coerper S, Beckert S, Witte MB, Konigsrainer A. Aging influences wound healing in patients with chronic lower extremity wounds treated in a specialized Wound Care Center. Wound Repair Regen. 2009 Jan-Feb;17(1):25-33. doi: 10.1111/j.1524-475X.2008.00438.x. PMID 19152648
- [Background] Richmond NA, Maderal AD, Vivas AC. Evidence-based management of common chronic lower extremity ulcers. Dermatol Ther. 2013 May-Jun;26(3):187-96. doi: 10.1111/dth.12051. PMID 23742279
- [Background] Frykberg RG, Banks J. Challenges in the Treatment of Chronic Wounds. Adv Wound Care (New Rochelle). 2015 Sep 1;4(9):560-582. doi: 10.1089/wound.2015.0635. PMID 26339534
- [Background] Edwards R, Harding KG. Bacteria and wound healing. Curr Opin Infect Dis. 2004 Apr;17(2):91-6. doi: 10.1097/00001432-200404000-00004. PMID 15021046
- [Background] Davis SC, Ricotti C, Cazzaniga A, Welsh E, Eaglstein WH, Mertz PM. Microscopic and physiologic evidence for biofilm-associated wound colonization in vivo. Wound Repair Regen. 2008 Jan-Feb;16(1):23-9. doi: 10.1111/j.1524-475X.2007.00303.x. PMID 18211576
- [Background] Game FL, Attinger C, Hartemann A, Hinchliffe RJ, Londahl M, Price PE, Jeffcoate WJ; International Working Group on the Diabetic Foot. IWGDF guidance on use of interventions to enhance the healing of chronic ulcers of the foot in diabetes. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:75-83. doi: 10.1002/dmrr.2700. No abstract available. PMID 26340818
- [Background] Phillips, P., Wolcott, R., Fletcher, J. & Schultz, G. S. Biofilms made easy. Wounds Int. 2010 1, 1-6.
- [Background] Herber OR, Schnepp W, Rieger MA. A systematic review on the impact of leg ulceration on patients' quality of life. Health Qual Life Outcomes. 2007 Jul 25;5:44. doi: 10.1186/1477-7525-5-44. PMID 17651490
- [Background] Niederauer MQ, Michalek JE, Armstrong DG. A Prospective, Randomized, Double-Blind Multicenter Study Comparing Continuous Diffusion of Oxygen Therapy to Sham Therapy in the Treatment of Diabetic Foot Ulcers. J Diabetes Sci Technol. 2017 Sep;11(5):883-891. doi: 10.1177/1932296817695574. Epub 2017 Feb 15. PMID 28654304